CLINICAL TRIAL: NCT03052595
Title: Multiple Sclerosis: The Role of Mitochondrial Dysfunction in Insulin Resistance
Brief Title: Multiple Sclerosis: The Role of Mitochondrial Dysfunction in IR Resistance
Acronym: MS-MIDY
Status: Completed | Type: Observational
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: Comenius University (Other)
Responsible Party: Principal Investigator, Adela Penesova, MD, PhD, Responsible Clinical Investigator, Slovak Academy of Sciences
Other Study IDs: APVV 15-0228
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis; Mitochondrial Alteration
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — MicroRNA, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SM: Patients with newly diagnosed multiple sclerosis undergo Oral glucose tolerance test to measure glucose and insulin concentrations after oral glucose load Patients undergo testing of autonomous nervous system function and testing of cognitive function (Stroop test)
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Testing of autonomous nervous system function; Diagnostic Test: Stroop test
- Control: Age, sex, Body Mass Index (BMI) matched healthy subjects undergo Oral glucose tolerance test to measure glucose and insulin concentrations after oral glucose load Healthy controls undergo testing of autonomous nervous system function and testing of cognitive function (Stroop test)
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Testing of autonomous nervous system function; Diagnostic Test: Stroop test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — Oral glucose tolerance test to measure glucose and insulin concentrations after oral glucose load
Diagnostic Test: Testing of autonomous nervous system function — Autonomous nervous system function will be assessed using a battery of tests (orthostasis, Valsalva manoeuvre, heart rate variability recording, blood hormone levels, ect.)
Diagnostic Test: Stroop test — Stroop test will be used to test cognitive function

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system (CNS) and is one of the most common neurological diseases, often leading to disability of the patients. The MS pathogenesis includes vascular and inflammatory components, however recently also the role of mitochondrial dysfunction being a hot topic in neurodegeneration.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system (CNS) and is one of the most common neurological diseases, often leading to disability of the patients. The MS pathogenesis includes vascular and inflammatory components, however recently also the role of mitochondrial dysfunction being a hot topic in neurodegeneration. Current project is based on previous project results, where the investigators of this project found signs of insulin resistance (IR) with hyperinsulinemia in patients with MS, which seem not to be related to chronic inflammation or low physical activity. Therefore aim of the present project is to elucidate impact of mitochondrial dysfunction in the pathogenesis of impaired insulin action and its role in the neurodegenerative process. To test the hypothesis, mitochondrial function, endothelial function, changes in membrane proteins and function of autonomic nervous system will be assessed. Those parameters will be measured non-invasively and in samples of blood, cerebrospinal fluid and skeletal muscle. MS patients will be examined at the time of diagnosis and after 12 months of treatment; healthy subjects will be used as controls. Elucidation of insulin resistance cause and the role of mitochondrial dysfunction in pathogenesis of disease is expected. Potential outcome of the project could be the answer, if pharmacological or non-pharmacological intervention might lead to improvement of mitochondrial function and therefore represent a new approach to prevent MS progression.

ELIGIBILITY:
Inclusion Criteria for MS patients:

* Age: 18-45 years
* Recent diagnosis of MS based on McDonald criteria
* Functional disability defined by the EDDS in the range of 2 to 6
* Patient demonstrates ability to successfully perform physical therapy exercises and procedures independently or with assistance of a caregiver

Exclusion Criteria:

* smoking, pregnancy, lactation, received a course of steroids (intravenous or oral) within 60 days of screening, diabetes, hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with newly diagnosed MS will be examined twice: immediately after the diagnosis confirmation and after at least 12 months of MS treatment
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2017-2019
  Insulin sensitivity indices calculated from plasma glucose and insulin concentrations during oral glucose tolerance test

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 2017-2020
  Expanded Disability Status Scale (EDSS) was developed for rating overall disability in MS. Patients are graded on the basis of presenting symptoms in eight different functional systems (FS), including pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, mental, and other functions. Scoring of the EDSS uses a 0 to 10, 20-step scale, with 0 equal to normal neurological function, 6.0 requires an assistive device for walking and 10.0 equal to death due to MS. The final score is based on grades obtained in the FS assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Viera Sevcikova, Ing, Study Chair — Biomedical Research Center of Slovak Academy of Sciences
Locations (1):
- Biomedical Center, Slovak Academy of Sciences, Institute of clinical and translational reasearch, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Imrich R, Vlcek M, Penesova A, Radikova Z, Havranova A, Sivakova M, Siarnik P, Kollar B, Sokolov T, Turcani P, Heckova E, Hangel G, Strasser B, Bogner W. Cardiac autonomic function in patients with early multiple sclerosis. Clin Auton Res. 2021 Aug;31(4):553-562. doi: 10.1007/s10286-021-00790-w. Epub 2021 Mar 4. PMID 33665745
- [Derived] Radikova Z, Penesova A, Vlcek M, Havranova A, Sivakova M, Siarnik P, Zitnanova I, Imrich R, Turcani P, Kollar B. Lipoprotein profiling in early multiple sclerosis patients: effect of chronic inflammation? Lipids Health Dis. 2020 Mar 17;19(1):49. doi: 10.1186/s12944-020-01221-x. PMID 32178676